CLINICAL TRIAL: NCT05757310
Title: A Pilot Study to Evaluate the Safety and Feasibility of Induction of Mixed Chimerism in Severe Aplastic Anemia Patients With COH-MC-17: A Non-Myeloablative/ Reduced-Intensity, Conditioning Regimen and CD4+ T-Cell-Depleted Haploidentical Hematopoietic Transplant
Brief Title: A Reduced-Intensity Conditioning Regimen (Cyclophosphamide, Pentostatin, Anti-thymocyte Globulin) Followed by Haploidentical Hematopoietic Stem Cell Transplant for the Treatment of Patients With Refractory or Recurrent Severe Aplastic Anemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23139; NCI-2022-10251 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23139 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-10; First posted 2023-03-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Severe Aplastic Anemia; Refractory Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Antilymphocyte Serum; Specimen Handling; Biopsy; Cyclophosphamide; Stem Cell Transplantation; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (conditioning, haploHCT) (Experimental): Patients receive cyclophosphamide PO and IV, pentostatin IV, anti-thymocyte globulin IV and undergo CD4+ T-cell depleted haploHCT on study. Patients also undergo bone marrow aspirate, bone marrow biopsy, and collection of blood samples at screening and follow-up.
  Interventions: Biological: Anti-Thymocyte Globulin; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspirate; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Procedure: Haploidentical Hematopoietic Cell Transplantation; Drug: Pentostatin; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATS
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspirate — Undergo bone marrow aspirate
  Other Names: Human Bone Marrow Aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cyclophosphamide — Given PO and IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Procedure: Haploidentical Hematopoietic Cell Transplantation — Undergo CD4+ T-cell depleted haploHCT
  Other Names: Haploidentical Stem Cell Transplantation; HLA-Haploidentical Hematopoietic Cell Transplantation; Stem Cell Transplantation, Haploidentical
Drug: Pentostatin — Given IV
  Other Names: (R)-3-(2-Deoxy-.beta.-D-erythro-pentofuranosyl)-3,6,7, 8-tetrahydroimidazo[4,5-d][1,3]diazepin-8-ol; 2'-Deoxycoformycin; CI-825; Co-Vidarabine; Covidarabine; DCF; Deoxycoformycin; Nipent; PD-81565; Pentostatine
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial evaluates the safety and feasibility of using a reduced-intensity regimen of cyclophosphamide, pentostatin, and anti-thymocyte globulin prior to a CD4+ T-cell depleted haploidentical hematopoietic cell transplant (haploHCT) for the treatment of patients with severe aplastic anemia that does not respond to treatment (refractory) or that has come back (recurrent). Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid. It may also lower the body's immune response. Pentostatin blocks a protein needed for cell growth. Anti-thymocyte globulin is an immunosuppressive drug can destroy immune cells known as T-cells. HaploHCT transfers blood-forming stem cells from a healthy partially-matched donor to a patient. Administering a regimen of cyclophosphamide, pentostatin, and anti-thymocyte globulin before haploHCT may help make room for the new, healthy cells and may reduce the risk of graft versus host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the infusion of CD4+ T-cell-depleted hematopoietic cells from a haploidentical donor, following a non-myeloablative/ reduced-intensity preparative regimen is safe in patients with severe aplastic anemia (SAA).

II. To determine the feasibility of producing an infusion ready CD4+ T-cell-depleted hematopoietic product, as assessed by:

IIa. Ability to meet the minimum required CD34+ cell dose, and; IIb. Ability to meet the CD4+ T-cell depletion product release requirements.

SECONDARY OBJECTIVES:

I. To evaluate toxicities including type, frequency, severity, attribution, time course, and duration. (Safety/tolerability) II. To summarize and evaluate hematologic (neutrophil and platelet) recovery, including marrow failure. (Safety/tolerability) III. To estimate the incidence of infection and infectious disease related complications at 100 days. (Safety/tolerability) IV. To estimate the incidence of SAA related complications. (Safety/tolerability) V. To estimate the cumulative incidence of non-relapse mortality at 100-days, 1-year and 2-years post hematopoietic stem-cell transplantation (HCT). (Safety/tolerability) VI. To estimate the cumulative incidence of acute graft versus host disease (GvHD) (grades: II-IV, III-IV) at 100-days and chronic GvHD (grades: any, moderate-severe) at 6-months, 1-year and 2-years post HCT. (Safety/tolerability) VII. To estimate the overall survival probability at 100-days, 1-year and 2-years post HCT. (Survival/relapse) VIII. To estimate the disease-free survival probability at 100-days, 1-year and 2-years post HCT. (Survival/relapse) IX. To estimate the event-free survival probability at 100-days, 1-year and 2-years post HCT. (Survival/relapse) X. To estimate the cumulative incidence of disease relapse at 100-days, 1-year and 2-years post HCT. (Survival/relapse) XI. To describe response as categorized by graft failure, persistent post-immunosuppressant (IS) mixed chimerism, persistent IS-dependent mixed chimerism, complete chimerism. (Chimerism) XII. To summarize/characterize patient chimerism (percent of donor total nucleated and donor lineage specific cells) over time. (Kinetics)

EXPLORATORY OBJECTIVES:

I. To describe the ratio of donor to recipient de novo thymic T cells over the course of 2 years within the peripheral blood compartment.

II. To describe the ratio of donor to recipient regulatory T cells and regulatory B cells over the course of 2 years within the peripheral blood and bone marrow compartments.

III. To describe the tolerance status of donor and host-type T cells over the course of 2 years within the peripheral blood compartment.

IV. To describe the T-cell repertoire of donor- and host-type T cells over the course of 2 years within the peripheral blood compartment.

V. To describe the bone marrow niche and peripheral blood cytokine profile over time.

VI. To describe bone marrow progenitor chimerism over time.

OUTLINE:

Patients receive cyclophosphamide orally (PO) and intravenously (IV), pentostatin IV, anti-thymocyte globulin IV and undergo CD4+ T-cell depleted haploHCT on study. Patients also undergo bone marrow aspirate, bone marrow biopsy, and collection of blood samples at screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* RECIPIENT: Documented informed consent of the participant.
* RECIPIENT: Age: >= 40 years but =< 75 years of age at time of enrollment.
* RECIPIENT: Failed at least one trial of immunosuppressive therapy (IST) by being refractory (persistence of severe cytopenia and fulfillment of SAA disease criteria at least 3 months after initial IST) or having relapsed (initial improvement of cytopenia after first-line IST but then a later return to fulfillment of SAA disease criteria when IST is decreased or ceased). IST could have included anti-thymocyte globulin (ATG) based regimens, calcineuPririn inhibitors and/or other higher dose therapy directed at the treatment of primary SAA.
* RECIPIENT: Karnofsky performance score >= 60%.
* RECIPIENT: Confirmed diagnosis of severe aplastic anemia as:

  * Bone marrow cellularity < 25% or marrow cellularity < 50% but with < 30% residual hematopoietic cells;
  * Two out of three of the following (in peripheral blood):

    * Neutrophils < 0.5 x 10^9/L;
    * Platelets < 20 x 10^9/L;
    * Reticulocyte count < 20 x 10^9/L (< 60 x 10^9/L using an automated analysis).
* RECIPIENT: No suitable fully matched related sibling donor (6/6 match for human leukocyte antigen [HLA]-A and B at intermediate or high resolution and DRbetaA1 at high resolution using deoxyribonucleic acid [DNA]-based typing) available.
* RECIPIENT: Available relative of the patient who is a haploidentical match, including biological parents, siblings or half siblings, children, uncles/aunts, first cousins, etc. Eligible haploidentical donors will have 2-4 mismatches if HLA-A, -B, -C, and -DRB1 typing is used; 2-5 mismatches if HLA-A, -B, -C, -DRB1, and -DQB1 typing is used; and 2-6 mismatches if HLA-A, -B, -C, -DRB1, -DQB1, and -DPB1 typing is used. A unidirectional mismatch in either the graft versus host or host versus graft direction is considered a mismatch. The donor and recipient must demonstrate that they are a full haplotype match by being identical at a minimum of one allele (at high resolution DNA-based typing) at the following genetic loci: HLA-A, -B, -C, and DRB1 if 8 allele typing is used; HLA-A, -B, -C, -DRB1, and -DQB1 if 10 allele typing is used; and HLA-A, -B, -C, -DRB1-, DQB1, and -DPB1 is 12 allele typing is used by the local center.
* RECIPIENT: Patient and/or legal guardian must sign informed consent for the hematopoietic stem cell transplantation (HSCT).
* RECIPIENT: The haplo donor and/or legal guardian must be able to sign informed consent documents.
* RECIPIENT: The potential haplo donor must be willing and able to donate bone marrow.
* RECIPIENT: The weight of the haplo donor must be >= 20 kg.
* RECIPIENT: Total bilirubin < 3.0 x the upper limit of normal (ULN) for age (patients who have been diagnosed with Gilbert's Disease are allowed to exceed this limit)
* RECIPIENT: Aspartate aminotransferase (AST) =< 5.0 x ULN.
* RECIPIENT: Alanine transaminase (ALT) =< 5.0 x ULN.
* RECIPIENT:

  * For patients >= 13.0 years of age at the time of enrollment: Creatinine clearance of >= 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula.
  * For patients < 13 years of age at enrollment: Glomerular filtration rate (GFR) estimated by the updated Schwartz formula > 90 mL/min/1.73 m^2. If the estimated GFR is < 90 mL/min/1.73m^2, then renal function must be measured by 24-hour creatinine clearance or nuclear GFR, and must be > 50mL/min/1.73m^2.
* RECIPIENT: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* RECIPIENT: Echocardiogram (ECHO) or multigated acquisition (MUGA): Left ventricular ejection fraction (LVEF) at rest >= 40%. For patients aged < 13 years, shortening fraction (SF) >= 26% by echocardiogram or MUGA may be substituted for LVEF.
* RECIPIENT:

  * For patients > 13.0 years of age: Diffusing capacity of the lung for carbon monoxide (DLCO) (corrected/adjusted for hemoglobin) > 40% and forced expiratory volume in 1 second (FEV1) > 50% predicted (without administration of bronchodilator) and forced vital capacity (FVC) > 50% predicted.
  * For patients < 13.0 years of age unable to perform pulmonary function tests (PFTs) due to age or developmental ability: (1) no evidence of dyspnea at rest and (2) no need for supplemental oxygen and (3) oxygen (O2) saturation > 92% on room air at sea level (with lower levels allowed at higher elevations per established center standard of care [e.g., Utah, 4,200 feet above sea level, does not give supplemental oxygen unless below 90%]).
* RECIPIENT: Seronegative for human immunodeficiency virus (HIV) antigen and antibody (Ag/Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR])

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed.
* RECIPIENT: Antibodies to donor red blood cell antigens including ABO and rhesus (Rh) meets institutional titer requirements.
* RECIPIENT: WOCBP or sexually active male: Agreement to use adequate contraception prior to study entry and 6 months post-CD4+ T-cell-depleted-HaploHCT.
* DONOR: Documented protocol-specific City of Hope (COH) informed consent per local, state and federal guidelines
* DONOR: Documented general institutional informed consent per local, state and federal guidelines.
* DONOR: Age: younger than 60 years.
* DONOR: Haplo donor selection is based on HLA typing and relationship to recipient.
* DONOR: When more than one donor is available, the donor with the lowest number of HLA allele mismatches will be chosen unless there is HLA cross-match incompatibility or a medical reason to select otherwise. In cases where there is more than one donor with the least degree of mismatch, donors will be selected based on the most favorable combination of HLA compatibility in cross-match testing and ABO compatibility. Prioritization is given to the lowest number of mismatches in the host-versus-graft (HVG) direction to minimize the risk of graft failure.
* DONOR: If there is more than one donor with the least amount of host-versus-graft (HVG) allele mismatches, the suggested prioritization in order of importance includes ABO compatibility, cytomegalovirus (CMV) status (use a sero-negative donor for a sero-negative recipient or use a sero-positive donor for a sero-positive recipient), younger age and lighter weight (this rule applies down to the age of 18, however, children may also be used as donors if appropriate), and sex of the donor (if all else is equal, males are preferred over nulliparous females over multiparous females).
* DONOR: Infectious disease screening performed within 30 days prior to stem cell collection and per federal guidelines and is:

  * Seronegative for HIV Ag, HIV 1+2 Ab, human T-lymphotropic virus (HTLV) I/II Ab, hepatitis B virus surface antigen (HBsAg), hepatitis B virus core antibody (HBcAb) (immunoglobulin M [IgM] and immunoglobulin G [IgG]), HCV Ab;
  * Negative RPR for syphilis.
* DONOR: WOCBP: Urine pregnancy testing performed within 7 days prior to stem cell mobilization
* DONOR: Is approved and completed evaluation per institutional guidelines.

Exclusion Criteria:

* RECIPIENT: Inherited and acquired (non-aplastic anemia) bone marrow failure syndromes such as Fanconi anemia must be ruled out according to center standards.
* RECIPIENT: Clonal cytogenetic abnormalities consistent with pre-myelodysplastic syndrome (pre-MDS) or MDS on marrow examination (e.g. Monosomy 7).
* RECIPIENT: Any somatic mutations (including TERT, TERC, DKC1, NOP10) other than PIG-A (PNH) or BCOR mutation.
* RECIPIENT: Diagnosis of myelodysplastic syndrome (MDS).
* RECIPIENT: Presence of anti-donor HLA antibodies (positive anti-donor HLA antibody is defined as a positive cross-match test of any titer by complement-dependent cytotoxicity or flow cytometric testing or the presence of anti-donor HLA antibody to the high expression loci HLA-A, B, C, DRB1, or DPB1 with mean fluorescence intensity [MFI] > 1000 by solid phase immunoassay).
* RECIPIENT: Prior allogeneic stem cell transplant.
* RECIPIENT: Prior solid organ transplant.
* RECIPIENT: Known life-threatening reaction (i.e., anaphylaxis) to Thymoglobulin (registered trademark) that would prohibit use for the patient as this study requires use of the Thymoglobulin (registered trademark) preparation of ATG.
* RECIPIENT: Uncontrolled bacterial, viral, or fungal infection at the time of enrollment. Uncontrolled is defined as currently taking medication and with progression or no clinical improvement on adequate medical treatment.
* RECIPIENT: Seropositive for the human immunodeficiency virus (HIV).
* RECIPIENT: Active hepatitis B or C determined by a detectable viral load of HBV or HCV.
* RECIPIENT: Female patients who are pregnant (per institutional practice) or breast-feeding.
* RECIPIENT: Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent > 5 years previously will be allowed. Cancer treated with curative intent =< 5 years previously will not be allowed unless approved by the protocol chairs and/or protocol officer.
* RECIPIENT: Alemtuzumab or ATG within 2 weeks of enrollment.
* RECIPIENT: Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* RECIPIENT: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).
* DONOR: Has undergone any transplantation (i.e. organ, stem cell, bone marrow, blood).
* DONOR: Receiving any investigational agents, or concurrent biological, chemotherapy, immunosuppression or radiation therapy.
* DONOR: Active infection.
* DONOR: Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis.
* DONOR: Factors which place the donor at increased risk for complications from leukapheresis or granulocyte colony-stimulating factor (G-CSF) therapy.
* DONOR: WOCBP: pregnant or =< 6 months breastfeeding.

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-06-18 (Estimated); Study Completion 2027-06-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From day -22 to day +100 or occurrence of unacceptable toxicity, whichever occurs first
  Toxicity will be graded according to the National Cancer Institute's-Common Terminology Criteria for Adverse Events version 5.0. Graft versus host disease (GVHD) specific toxicities will be defined per 1994 Keystone Consensus Criteria. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study regimen and reversibility or outcome. This will include infectious disease related complications and autoimmune disease related complications. Cumulative incidence curves will be used for time to event variables with competing risks events such as acute GVHD or chronic GVHD. Point estimates and 90% confidence intervals will be used.
Ability to meet CD4+ T-cell depleted product release requirements (feasibility) | Up to 3 years
  The feasibility of producing an infusion ready CD4+ T-cell-depleted hematopoietic product will be assessed by the ability to meet product release requirements. Product release requirements include the following: (1) CD34+ cells: Post-processing CD34+ cell target of 7.5-13.0 x 106 cells/kg of recipient body weight; (2) CD4+ T-cell depletion: >= 97% of CD4+ T-cells in the the hematopoietic cell product for manufacturing; (3) Sterility (e.g. endotoxin and gram staining). Descriptive statistics will be used to characterize feasibility.
Ability to meet minimum required cell dose (feasibility) | Up to 3 years
  The feasibility of producing an infusion ready CD4+ T-cell-depleted hematopoietic product will be assessed by the ability to meet minimum required cell doses. This outcome will be evaluated using the following: (1) CD34+ collected (per day of apheresis); (2) CD34+ recovery: % CD34+ cells recovered from the CD34+ cell number in the product being manufactured (pre-CD4+ T cell depletion); (3) Cell dose: pooled and back up product; (4) Cell dose adequate given recipient's body weight plus the required pre-processed back-up set aside (yes/no); (5) Number (median, range) of apheresis; (6) % CD4+ T-cell depletion; (7) reason for not meeting product release requirements. Descriptive statistics will be used to characterize feasibility.

SECONDARY OUTCOMES:
Incidence of adverse events of grade 3 or higher | Up to 3 years
Incidence of infection | Up to 3 years
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any.
Time to neutrophil recovery | From the date of CD4+ T-cell-depleted product infusion to the first of three consecutive days of absolute neutrophil count (ANC) >= 500/mm^3 and ANC >= 1000/mm^3, assessed up to 3 years
Time to platelet recovery | Time to the first day of the first of three consecutive laboratory values when the platelet count is >= 20,000/mm^3 and 100,000/mm^3 without a platelet transfusion in the previous seven, assessed up to 3 years
Marrow failure | Up to 28 days post transplant for primary graft failure or after initial engraftment for secondary graft failure, assessed up to 3 years
  Defined as primary graft failure: failure to achieve a sustained neutrophil count of >= 500/ mm^3 in the absence of disease relapse by 28 days or secondary graft failure: a decline in the neutrophil count to less than 500/ mm^3 after initial engraftment, which was unrelated to infection, medications, or disease relapse.
Cumulative incidence of non-relapse mortality (NRM) | From enrollment until non-disease related death or last follow up and from date of CD4+ T-cell-depleted product infusion, assessed up to 3 years
  NRM is defined as death occurring in a patient from causes other than disease relapse; relapse is a competing event. Cumulative incidence curves will be used for time to event variables with competing risks events. Point estimates and 90% confidence intervals will be used.
Cumulative incidence of acute GvHD (II-IV and III-IV) | From day 0 through day +100 post-transplant
  Acute GvHD is graded according to the Keystone Consensus Criteria. The first day of acute GvHD onset at a certain grade will be used to calculate cumulative incidence curves; death is a competing event. Cumulative incidence curves will be used for time to event variables with competing risks events. Point estimates and 90% confidence intervals will be used.
Cumulative incidence of chronic GvHD (any and moderate-severe) | From day +100 to +2 years post-transplant
  Chronic GvHD is graded according to the 2014 NIH Consensus Criteria. The first day of chronic GvHD onset at a certain grade will be used to calculate cumulative incidence curves; disease recurrence or death is a competing event. Cumulative incidence curves will be used for time to event variables with competing risks events. Point estimates and 90% confidence intervals will be used.
Overall survival | Time from enrollment to death, assessed up to 3 years
  Patients are considered a failure for this endpoint if they die, regardless of cause of death. Overall survival will be censored at last follow-up if patients are known to be alive. Kaplan-Meier curves will be used for time to event variables.
Cumulative incidence of relapse | Time from enrollment/infusion of depleted hematopoietic product to first observation of disease relapse, assessed up to 3 years
  Disease relapse is defined as a decline in the neutrophil count to less than 500/ mm^3 after initial engraftment, which was unrelated to infection, medications, or other causes. Death without disease recurrence will be a competing risk event. Time to disease recurrence will be censored at the last disease assessment of patients remain alive and free of disease recurrence.
Disease-free survival (DFS) | Time from enrollment/ infusion of CD4+ T-cell-depleted hematopoietic product to relapse, therapy for hemoglobinopathy, death from any cause, assessed up to 3 years
  Patients are considered a failure for this endpoint if they relapse or die, regardless of cause of death. DFS will be censored at last follow-up if patients are alive and free of disease. Kaplan-Meier curves will be used for time to event variables.
Event-free survival (EFS) | Time from enrollment/infusion of CD4+ T-cell product to any of the following events (whichever occurs first): therapy for hemoglobinopathy, primary/secondary graft failure, acute GvHD, chronic GvHD, death from any cause, assessed up to 3 years
  EFS will be censored at last follow-up if patients are free of any above-mentioned events. Kaplan-Meier curves will be used for time to event variables.
Chimerism | Up to 2 years
  Persistent IS-dependent mixed chimerism: Between 10% and 94% donor chimerism at two years post-transplant and on IS. Complete chimerism: >94% donor chimerism at two years post-transplant. Primary donor graft failure: Defined as < 10 % donor chimerism by day +30 post-transplant.. Secondary donor graft failure: Defined as < 10 % donor chimerism beyond day +30 in patients with prior documentation of >= 10% donor cells by day +30. Failure is based on two separate measurements obtained at least 2 weeks apart. Line charts or scatterplots will be used for changes of endpoints over time such as chimerism.
Kinetics | At 7, 15, 30, 60, 100, 180 days and 1, 1.5, and 2 years post-transplant
  Will evaluate T-cells: CD3, CD4, CD8, B-cells: CD19, natural killer cells: CD56, monocytes: CD14, granulocytes: CD15, total nucleated cells. Line charts or scatterplots will be used for changes of endpoints over time.

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States